CLINICAL TRIAL: NCT04485052
Title: A Phase Ib Study Evaluating the Safety and Efficacy of IBI188 in Combination With Demethylating Agents in Subjects With Acute Myeloid Leukemia
Brief Title: Efficacy and Safety Evaluation of IBI188 in Combination With Demethylating Agents in Treatment of Patients With Acute Myeloid Leukemia
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pause for changes in development strategies
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188B201
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI188+azacitidine (Experimental): 1L unfit AML receive IBI188 every week by intravenous(IV) and azacitidine daily in Day 1-7 of each four weeks(Q4W) by subcutaneous(IH)
  Interventions: Drug: IBI188; Drug: Azacitidine
- IBI188+decitabine (Experimental): R/R AML receive IBI188 every week by intravenous(IV) and decitabine daily in Day 1-10 of each four weeks(Q4W) by subcutaneous(IH)
  Interventions: Drug: IBI188; Drug: Decitabine

INTERVENTIONS:
Drug: IBI188 — anti-CD47 Monoclonal antibody
Drug: Azacitidine — Demethylation drugs
  Arms: IBI188+azacitidine
Drug: Decitabine — Demethylation drugs
  Arms: IBI188+decitabine

SUMMARY:
The study is to evaluate safety, tolerability and composite CR of IBI188 plus Demethylating Agents in acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

1. AML patients diagnosed according to WHO AML diagnostic criteria in 2016 (except M3-type and BCR-ABL positive AML).
2. Relapsed// refractory AML( ≥18 ys) or newly diagnosed elderly AML unfit for intensive chemotherapy( ≥60 ys).
3. Age ≥18 years old, gender not limited.
4. ECOG score of 0-2.
5. Adequate organ function.

Exclusion Criteria:

1. Acute promyelocytic leukemia, myeloid sarcoma, acute heterozygous leukemia, CMML(accelerated phase and blast phase).
2. A history of myeloproliferative diseases (including myelofibrosis, primary thrombocytosis, and true red) Cytosis, chronic myelocytic leukemia) or acute myeloid white blood with BCR-ABL1 translocation Patients.
3. Major surgery and vaccine treatment within 4 weeks.
4. Uncontrolled concurrent diseases.
5. Pregnant or breastfeeding female subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite complete rate | 24 weeks
  Composite CR including complete remission rate and morphologic complete remission with incomplete blood count recovery

SECONDARY OUTCOMES:
Cytogenetic CR | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China